CLINICAL TRIAL: NCT02260570
Title: Remediation of Impaired Self-Regulation in Patients With Mild TBI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Berkeley (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D0825-I; 1I01RX000825-01 (NIH)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mild Traumatic Brain Injury
Keywords: concussion; MRI; memory; tolcapone; post-traumatic stress disorder
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic | interventions — Tolcapone

STUDY DESIGN:
Intervention Model Description: In this study, subjects received either tolcapone or placebo in randomized, double-blind, counterbalanced fashion. The study is a single arm study in which all subjects receive both tolcapone and placebo, but to comply with clinical trial reporting requirements, it is listed here as a two arm study: one arm for subjects who received tolcapone first, and one arm for subjects who received placebo first. Because baseline dopamine levels can vary substantially between individuals, this grouping by sequence rather than by drug condition retains the within-subject information necessary for subsequent analyses. The alternative (grouping by tolcapone or placebo) loses this within-subject information.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional MRI Arm 1: Tolcapone first, then placebo (Experimental): This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Subjects have been divided into two arms based on the order in which they received the drug intervention. Because baseline dopamine levels can vary substantially between individuals, this grouping by sequence rather than by drug condition retains the within-subject information necessary for subsequent analyses.
  Interventions: Drug: Tolcapone; Drug: Placebo
- Functional MRI Arm 2: Placebo first, then tolcapone (Experimental): This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Subjects have been divided into two arms based on the order in which they received the drug intervention. Because baseline dopamine levels can vary substantially between individuals, this grouping by sequence rather than by drug condition retains the within-subject information necessary for subsequent analyses.
  Interventions: Drug: Tolcapone; Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — COMT Inhibitor
  Other Names: Tasmar
Drug: Placebo — A pill that contains no active ingredient

SUMMARY:
The ability to regulate impulses enables us to plan for the future, to maintain focus in the face of distractions (i.e. to encode memories), and to manage emotions. This self regulation can be compromised in individuals who have a history of mild traumatic brain injury and co-occurring disorders. In this study the investigators are using functional MRI scanning to understand how memory and self regulation are expressed in the brains of people with a history of mild traumatic brain injury. The investigators are also testing whether the medication tolcapone may improve memory and self regulation.

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled, crossover cognitive neuroscience study, the investigators are evaluating whether the catechol-O-methyltransferase (COMT) inhibitor tolcapone impacts memory and self regulation, as measured both behaviorally (via cognitive testing) and neurophysiologically (via functional MRI).

ELIGIBILITY:
Inclusion Criteria:

* Veteran ages 18-50 and in general good health;
* Able to read English at a 6th grade level;
* Able to provide written informed consent;
* Normal or corrected to normal visual acuity;
* Stable doses of all medications (2 weeks or greater);
* History of mild traumatic brain injury greater than 6 months prior to participation

Exclusion Criteria:

* Contraindications to magnetic resonance imaging (MRI) scanning;
* Inability to complete basic fMRI requirements;
* History of brain surgery or penetrating brain injury;
* Uncontrolled blood pressure (low or high);
* Contraindications to tolcapone use;
* Use of medications or drugs with dopamine-related actions within 30 days;
* Active substance abuse or dependence;
* Clinically severe medical illness requiring treatment;
* History of psychiatric hospitalization (past 1 year) or suicide attempt (past 5 years);
* Seizures greater than 4 weeks after traumatic brain injury (TBI) event or seizures requiring active treatment;
* History of brain tumor, stroke, Alzheimer's disease, aneurysm rupture, or multiple sclerosis;
* History of schizophrenia, attention deficit hyperactivity disorder (ADHD) or psychiatric diagnosis EXCEPT depression or post-traumatic stress disorder (PTSD)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Kayser, MD PhD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Westphal AJ, Ballard ME, Rodriguez N, Vega TA, D'Esposito M, Kayser AS. Working memory, cortical dopamine tone, and frontoparietal brain recruitment in post-traumatic stress disorder: a randomized controlled trial. Transl Psychiatry. 2021 Jul 12;11(1):389. doi: 10.1038/s41398-021-01512-6. PMID 34253715
- See also: Reference + link to the published open-access manuscript — https://pubmed.ncbi.nlm.nih.gov/34253715/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects participated in a single-arm study in which all subjects received tolcapone and placebo in randomized, counterbalanced, crossover fashion. Because baseline dopamine levels can differ substantially between individuals, each subject serves as their own control. As a result, compiling data for a "tolcapone" arm and a "placebo" arm is not preferred, as such a grouping ignores the within-subject comparison. Instead, subjects are grouped "per sequence".
Pre-assignment Details: Subjects were screened based on inclusion and exclusion criteria. Only eligible subjects were assigned to a study arm. 55 subjects provided informed consent to participate in screening and study procedures, but after the screening visit, only 35 subjects were determined to be eligible to proceed to study arm assignment.
Groups:
- Functional MRI Arm 1: Tolcapone First, Then Placebo; Functional MRI Arm 2: Placebo First, Then Tolcapone: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. For reporting purposes, subjects have been divided into two arms based on the order in which they received the drug intervention. Because baseline dopamine levels can vary substantially between individuals, this grouping retains the within-subject information necessary for subsequent analyses.
  Tolcapone: COMT Inhibitor
  Placebo: A pill that contains no active ingredient
Period: Overall Study
Arm/Group | Functional MRI Arm 1: Tolcapone First, Then Placebo | Functional MRI Arm 2: Placebo First, Then Tolcapone
Started | 18 | 17
Completed | 15 | 15
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: The total number of subjects reflects the number who completed all study procedures.
Groups:
- Baseline Data for All Subjects: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Baseline information was obtained across the entire group, not per arm
  Tolcapone: COMT Inhibitor
  Placebo: A pill that contains no active ingredient
Arm/Group | Baseline Data for All Subjects
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — The mean and standard deviation reported for age reflect the total number of completed subjects.
  years | 35.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 3
  Unknown or Not Reported | 0
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — The mean and standard deviation reported for the CAPS-5 reflect the total number of subjects who completed all study procedures. (CAPS-5 scores 0-68, where scores of 31-33 or higher suggest the need for PTSD treatment).
  units on a scale | 25.4 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Brain Signal Measured Using Functional MRI.
Description: Functional MRI measures blood flow changes. Blood Oxygen Level Dependent (BOLD) signals provide an indirect unitless measure of brain activity typically described as a percentage. However, because fMRI data sets are large (> 10,000 comparisons), analysis packages present results as F statistics or similar measures for individual voxels across the brain. Thus, no single mean or median value describes the 3-way interaction between drug (tolcapone minus placebo), stimulus emotion (neutral versus anxious), and CAPS-score with degrees of freedom = [1,1,60]. Because each subject serves as his/her own control, drug results are also intrinsically paired -- i.e. data are presented for participants as tolcapone minus placebo results within subject. The data values below represent the number of above-threshold, neighboring voxels in the largest clusters of voxels in the brain for the patient group as a whole, not separately for each participant.
Time Frame: Approximately 60-240 minutes following tolcapone/placebo administration
Population: Using the Analysis of Functional Neuroimaging (AFNI) package, we implemented a 3-way ANOVA for the interaction between drug (tolcapone minus placebo), stimulus emotion (neutral versus anxious), and CAPS score. In the summary analysis below, the number of suprathreshold voxels below represents 2.65mm3 isotropic voxels in the left frontal pole and right inferior gyrus, respectively. It is a count, not a mean, and the fMRI package does *not* provide bootstrapped ranges for suprathreshold voxels.
Measure: Number; unit: voxels
Groups:
- Tolcapone: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Because baseline dopamine levels can vary substantially between individuals -- i.e. there is high inter-subject variability in baseline dopamine levels -- the primary outcome measures rely upon *within-subject* comparisons of tolcapone versus placebo, not across-group comparisons.
  Tolcapone: COMT Inhibitor
- Placebo: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Because baseline dopamine levels can vary substantially between individuals -- i.e. there is high inter-subject variability in baseline dopamine levels -- the primary outcome measures rely upon *within-subject* comparisons of tolcapone versus placebo, not across-group comparisons.
  Placebo: A pill that contains no active ingredient
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 30 | 30
voxels | 270 | 111
Statistical Analysis 1: Comparison: Tolcapone vs Placebo; Test type: Superiority; p < 0.0001, ANOVA — This p-value is adjusted for multiple comparisons; F(1,1,60) = 24.1, p < 0.0001, adjusted r^2 = 0.275; F value = 24.1

2. Primary Outcome: Performance on Cognitive Testing
Description: Tasks to assess cognition were performed while subjects are scanned. Signal detection theory (SDT) assesses the ability of subjects to accurately recall working memory memoranda. In SDT, the sensitivity index d' results from subtracting the normalized false alarm rate from the normalized hit rate; thus, higher values of d' indicate better working memory performance.
  Here we evaluate the interaction with respect to d' between drug condition (tolcapone minus placebo) and Post-Traumatic Stress Disorder severity as measured by the total score on the *Clinician Administered PTSD Scale*, or CAPS. Total CAPS scores range from 0 to 80, with higher scores indicating greater PTSD severity. Because each subject serves as his/her own control, drug results for behavior are intrinsically paired -- i.e. data are presented for participants as tolcapone minus placebo results, as prespecified in the statistical analysis plan.
Time Frame: Approximately 60-240 minutes following tolcapone/placebo administration
Population: The population of 30 subjects evaluated in this single arm study is described elsewhere in this record. Here we used a 2-way ANOVA to evaluate the interaction between drug (tolcapone minus placebo) and CAPS-score with respect to the working memory performance measure d', taken from signal detection theory and based upon the hit rate and false alarm rate.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 25.4 [0 to 68] | 25.4 [0 to 68]
Statistical Analysis 1: Comparison: Tolcapone vs Placebo; Test type: Superiority; p = 0.0184, ANOVA — This p-value is adjusted for multiple comparisons; F(1,30) = 6.23, p = 0.0184, adjusted r^2 = 0.144; F value = 6.23

ADVERSE EVENTS:
Time Frame: In this study, subjects were administered tolcapone and placebo once each on the two study days. Adverse event data were recorded for the two days in which subjects participated.
Description: Adverse events were defined as per clinicaltrials.gov.
Groups:
- Functional MRI Arm 1: Tolcapone: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion.
  Tolcapone: a COMT Inhibitor
- Functional MRI Arm 2: Placebo: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion.
  Placebo first: A pill that contains no active ingredient
Arm/Group | Functional MRI Arm 1: Tolcapone | Functional MRI Arm 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
For additional details, including results discussion, please see the primary resulting open-access publication:

Westphal AJ, Ballard ME, Rodriguez N, Vega TA, D'Esposito M, Kayser AS. Enhancing prefrontal dopamine tone improves working memory and recruits frontoparietal brain regions in individuals with post-traumatic stress disorder. Translational Psychiatry, 11(1): 389.

This reference is also included in the References module of the Protocol section for this ClinitalTrials.gov record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT02260570/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT02260570/ICF_001.pdf